CLINICAL TRIAL: NCT05066854
Title: INterest of the Negative Predictive Value of Integrons in Choosing a Narrow-spectrum Empirical anTibiotic Treatment vs Usual Empirical Antibiotic Treatment for Urinary Tract infectionS in the PEDiatric Emergency Department
Acronym: INVICTUS PED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI20_0029 (INVICTUS PED)
Record Dates: First submitted 2021-09-16; First posted 2021-10-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Urinary Tract Infections in Children
Keywords: empirical antibiotic treatment; biomarker; urinary tract infection; antibiotic resistance; pediatric emergency department
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integron research (Experimental): Empirical antibiotic treatment chosen based on the results of the integron search:
  * when PCR is negative, patients will receive SXT (30 mg/kg/j of sulfamethoxazole and 6 mg/kg/j of trimethoprim)
  * when PCR is positive or uninterpretable for integrons, patients will receive an empirical antibiotic treatment based on the usual practice of each center according to the GPIP guidelines.
  Interventions: Procedure: integron research
- Usual practice (Other): Empirical antibiotic treatment based on the usual practice of each center according to the GPIG guidelines.
  Interventions: Procedure: usual practice

INTERVENTIONS:
Procedure: integron research — Patients with suspected UTI with fever will be screened at their admission to the pediatric ED.
  Urine samples will be sent to the laboratory for culture and integron PCR according to routine practice.
  Results of the integron search will be given to the investigator. Patients in the experimental group with a positive or uninterpretable PCR will also receive an empirical antibiotic treatment based on the usual practice of each center according to the GPIP guidelines.
  Patients in the experimental group with a negative PCR will receive a treatment with SXT at the recommended dose.
  Arms: Integron research
Procedure: usual practice — Patients with suspected UTI with fever will be screened at their admission to the pediatric ED.
  Patients in the control group will receive an empirical antibiotic treatment based on the usual practice of each center according to the GPIP guidelines.
  Arms: Usual practice

SUMMARY:
INVICTUS PED primary objective is to show the non-inferiority of an empirical antibiotic therapeutic management guided by the early detection of integrons in the urine, compared to a usual empirical antibiotic treatment, for the recovery of children admitted to the pediatric emergency department (ED) with a non-severe urinary tract infection (UTI) with fever

DETAILED DESCRIPTION:
Urinary tract infections with fever are common in children and require primary health care management. Because of the risk of immediate evolution to a systemic infection with long-term renal scars, empirical antibiotic treatment is recommended. The French Group for Pediatric Infectious Diseases (GPIP) recommends the use of third-generation cephalosporins (3GC) targeting enterobacteria, which are mainly involved in UTI and increasingly resistant to antibiotics through the production of extended-spectrum β-lactamases. However, use of 3GC is a well-known risk factor for resistant germs selection and one of the main guideline to fight antibiotic resistance, which is an important public health issue, is to reduce their use. Integrons are genetic elements involved in the spread of antibiotic resistance in enterobacteria. Preliminary studies showed that integron search using polymerase chain reaction (PCR) directly on urine samples had a great NPV (>98%) for trimethoprim-sulfamethoxazole (SXT). The hypothesis is that, in children presenting to the pediatric ED with non-severe UTI with fever, absence of integron in their urine could allow prescribing an empirical antibiotic treatment with SXT without decreasing the chance of recovery, thus decreasing the use of 3GC.

Two strategies is compare: i) In the control group: empirical antibiotic treatment according to the usual practice of each center, in line with the GPIP guidelines, ii) in the experimental group: empirical antibiotic treatment chosen depending on the results of the integron search with PCR. When PCR is positive, treatment according to usual practice; when PCR is negative, treatment with SXT.

Two follow-up visits, by phone, will be planned: at H48 (+ 24h), when the empirical antibiotic treatment is assessed based on the urine culture and antimicrobial susceptibility test (AST) results, and on D30 (+/- 2 days) at the end of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children above 3 months old and under 18 years old
* Consultation in a participating pediatric emergency department
* Suspicion of UTI with fever (Fever ≥ 38°C and urine dipstick test positive for leukocytes and/or nitrites)
* First episode of UTI with fever
* Written informed consent of the holders of parental authority
* Affiliated to Social Security

Exclusion Criteria:

* Criteria of severity:

  * Severe infection with severe sepsis or septic shock
  * Dehydration ≥ 10%
  * Fever ≥ 38°C > 4 days (96h)
  * Indication of surgical or interventional drainage
* Complication risk factors:

  * Any anatomic or functional defect of the urinary tract (other than low-grade VUR and calyceal dilation < 10 mm)
  * Repetition of UTI with fever ≤ than 6 months since the previous episode
  * Repetition of UTI with fever and anatomic or functional defect of the urinary tract
  * Pregnancy
  * Severely immunocompromised patient
  * Severe chronic renal failure defined as a clearance < 30 mL/min/1.73 m2
  * Severe liver failure
* 3GC allergy
* Contra-indication to SXT:

  * G6PD deficiency
  * Treatment with methotrexate
  * Allergy to sulfonamide
* Antibiotic treatment within 48h before admission
* Empirical antibiotic treatment not recommended

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Recovery | Day 30
  Recovery defined as, apyrexia obtained within less than 72h and no persistence or repetition of UTI with fever and no change of empirical antibiotic therapy required because of resistance and no treatment interruption for adverse effects

SECONDARY OUTCOMES:
patients treated | Day 30
  Number of patients treated with 3GC in both groups, during the participation of each patient
Duration treatment | Day 30
  Duration of treatment with 3GC in both groups for patient treated, during the participation of each patient
Antibiotic treatment changes | Hour 48
  In both groups, description of antibiotic treatment changes based on the AST results, according to 4 criteria:
  * Change because of resistance
  * Narrowing of the antibiotic spectrum
  * Interruption because the diagnosis of UTI was ruled out
  * Antibiotics used
Adaptation of antibiotherapy with the AST result | Hour 48
  Proportion of patients in both groups for whom empirical antibiotic treatment was adapted to the AST results and did not require any change (because of resistance, or to narrow the antibiotic spectrum)
Resistance of enterobacteria | Hour 48
  In the study population, percentage of resistance of enterobacteria to the different antibiotic classes
Predictive values of the integrons | Hour 48
  Negative and positive predictive values of the integrons depending on the main antibiotic classes used in the experimental group.
Apyrexia | Hour 48
  Time to apyrexia from the start of the antibiotic therapy compared between both groups.
Early repetition of urinary tract infection | Day 30
  Proportion of early repetition of urinary tract infection with fever in both groups.
Treatment interruption for adverse effects | Day 30
  Proportion of treatment interruption for adverse effects in both groups.
Time spent in the pediatric emergency department | Day 30
  Time spent in the pediatric emergency department in both groups

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Bordeaux university Hospital, Bordeaux
  - Limoges university Hospital, Limoges
  - Montpellier university Hospital, Montpellier
  - Toulouse university Hospital, Toulouse